CLINICAL TRIAL: NCT03948685
Title: Carvedilol SR Study for Biomarkers From Blood and Urine and Safety of in Patients With Heart Failure With Preserved Ejection Fraction : a Prospective, Randomized, Double Blind, Placebo-controlled, Multicenter, Pilot Trial (CAYMUS-HFpEF)
Brief Title: Carvedilol SR Study for Biomarkers From Blood and Urine and Safety of in Patients With Heart Failure With Preserved Ejection Fraction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-1061
Record Dates: First submitted 2019-05-03; First posted 2019-05-14 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Intervention Model Description: Carvedilol SR vs. Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol SR (Experimental): Carvedilol SR 8mg, 16mg, 32mg
  Interventions: Drug: Carvedilol SR
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol SR — blood pressure, heart rate based titrated carvedilol SR for 24 weeks
  Arms: Carvedilol SR
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Beta blockers have been used to reduce the mortality and heart failure rehospitalization in heart failure with reduced ejection fraction (HFrEF) patients in addition to ACEI/ARB, MRA, ivabradine and ARNI. However, the effective and safe medical therapy is not well established in heart failure with preserved ejection fraction (HFpEF) yet. Recent meta-analysis showed that beta blockers may also be beneficial for reducing the mortality and heart failure rehospitalization in HFpEF like HFrEF. However, the clinical effect and safety of carvedilol have been largely unknown in HFpEF. Therefore, CAYMUS HFpEF is the exploratory study to assess the change of surrogate markers (NTproBNP, hsTn) when treated with carvedilol SR vs. placebo in HFpEF patients

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedure
2. Male or female, aged ≥ 19 years
3. Patients with chronic HF (Chronic Heart Failure) NYHA (New York Heart Association classification) class II-IV and preserved EF (Ejection Fraction)(LVEF (Left Ventricular Ejection Fraction) > 40 %) and elevated NT-proBNP (N-terminal of the prohormone brain natriuretic peptide) > 200 pg/ml for patients without AF, OR > 600 pg/ml for patients with AF, analysed at the Central laboratory at Visit 1
4. Structural heart disease within 6 months prior to Visit 1 using echocardiagraphy

Exclusion Criteria:

1. Myocardial infarction, coronary artery bypass graft surgery or other major cardiovascular surgery, stroke or TIA (Transient Ischaemic Attack) in past 90 days prior to Visit 1
2. Contraindication to beta blocker
3. Heart transplant recipient or listed for heart transplant
4. Hospitalization plan for PCI, coronary artery bypass graft surgery, other cardiac invasive interventions (e.g. catheter ablation, pacemaker, CRT, ICD implantation)
5. Acute decompensated HF (Heart Failure)
6. Symptomatic hypotension or systolic blood pressure < 100 mmHg)
7. Patients with CrCl < 30 ml/min using creatinine-based CKD-EPI equations
8. Elevated liver enzymes (3 times over upper reference limit) or liver cirrhosis
9. Symptomatic bradycardia or heart rate < 60/min
10. Allergy, adverse drug reaction, hypersensitivity to carvedilol
11. Life expectancy < 6 months (e.g. metastatic malignancy)
12. Pregnancy, or women of childbearing age

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
The Maximum NT-proBNP value change after Drug(Carvedilol SR or Placebo) administration. | Baseline
  The maximum NT-proBNP value change at baseline.
The Maximum NT-proBNP value change after Drug(Carvedilol SR or Placebo) administration. | 8 weeks
  The maximum NT-proBNP value change from baseline to 8 weeks.
The Maximum NT-proBNP value change after Drug(Carvedilol SR or Placebo) administration. | 24 weeks
  The maximum NT-proBNP value change from baseline to End of trial(24weeks).

SECONDARY OUTCOMES:
The changes of maximum surrogate markers values(hsTn, hsCRP, sST2, Galectine-3, IGFBP7, Neprilysin, D-dimer, MMP-2, Cystatin C, NAG, NGAL, KIM-1, BUN, Creatinine, Chloride, Na, K, PICP and spondin-1) after Drug(Carvedilol SR or Placebo) administration. | Baseline
  the change of surrogate markers(hsTn, hsCRP etc) at baseline.
The changes of maximum surrogate markers values(hsTn, hsCRP, sST2, Galectine-3, IGFBP7, Neprilysin, D-dimer, MMP-2, Cystatin C, NAG, NGAL, KIM-1, BUN, Creatinine, Chloride, Na, K, PICP and spondin-1) after Drug(Carvedilol SR or Placebo) administration. | 8 weeks
  the change of surrogate markers(hsTn, hsCRP etc) after 8 weeks.
The changes of maximum surrogate markers values(hsTn, hsCRP, sST2, Galectine-3, IGFBP7, Neprilysin, D-dimer, MMP-2, Cystatin C, NAG, NGAL, KIM-1, BUN, Creatinine, Chloride, Na, K, PICP and spondin-1) after Drug(Carvedilol SR or Placebo) administration. | 16 weeks
  the change of surrogate markers(hsTn, hsCRP etc) after 16 weeks.
The changes of maximum surrogate markers values(hsTn, hsCRP, sST2, Galectine-3, IGFBP7, Neprilysin, D-dimer, MMP-2, Cystatin C, NAG, NGAL, KIM-1, BUN, Creatinine, Chloride, Na, K, PICP and spondin-1) after Drug(Carvedilol SR or Placebo) administration. | 24 weeks
  the change of surrogate markers(hsTn, hsCRP etc) from baseline to end of trial(24 weeks)
The change in degree of dyspnea using VAS questionnaire | Baseline
  the change of dyspnea at baseline.
The change in degree of dyspnea using VAS questionnaire | 8 weeks
  the change of dyspnea after 8 weeks.
The change in degree of dyspnea using VAS questionnaire | 16 weeks
  the change of dyspnea after 16 weeks.
The change in degree of dyspnea using VAS questionnaire | 24 weeks
  the change of dyspnea from baseline to end of trial(24 weeks)
the change of body weight | Baseline
  the change of body weight at baseline.
the change of body weight | 8 weeks
  the change of body weight after 8 weeks.
the change of body weight | 16 weeks
  the change of body weight after 16 weeks.
the change of body weight | 24 weeks
  the change of body weight from baseline to end of trial(24 weeks)
the frequency of symptomatic hypotension, symptomatic bradycardia and AV block above 2nd degree | Baseline
  the frequency of symptomatic hypotension, symptomatic bradycardia and AV block above 2nd degree during the tiral
the frequency of symptomatic hypotension, symptomatic bradycardia and AV block above 2nd degree | 8 weeks
  the frequency of symptomatic hypotension, symptomatic bradycardia and AV block above 2nd degree during the tiral
the frequency of symptomatic hypotension, symptomatic bradycardia and AV block above 2nd degree | 16 weeks
  the frequency of symptomatic hypotension, symptomatic bradycardia and AV block above 2nd degree during the tiral
the frequency of symptomatic hypotension, symptomatic bradycardia and AV block above 2nd degree | 24 weeks
  the frequency of symptomatic hypotension, symptomatic bradycardia and AV block above 2nd degree during the tiral
the frequency of hypo/hyperkalemia and worsening kidney function | Baseline
  the frequency of hypo/hyperkalemia and worsening kidney function during the trial
the frequency of hypo/hyperkalemia and worsening kidney function | 8 weeks
  the frequency of hypo/hyperkalemia and worsening kidney function during the trial
the frequency of hypo/hyperkalemia and worsening kidney function | 16 weeks
  the frequency of hypo/hyperkalemia and worsening kidney function during the trial
the frequency of hypo/hyperkalemia and worsening kidney function | 24 weeks
  the frequency of hypo/hyperkalemia and worsening kidney function during the trial
all-cause hospitalization & mortality | Baseline
  all-cause hospitalization & mortality during the trial
all-cause hospitalization & mortality | 8 weeks
  all-cause hospitalization & mortality during the trial
all-cause hospitalization & mortality | 16 weeks
  all-cause hospitalization & mortality during the trial
all-cause hospitalization & mortality | 24 weeks
  all-cause hospitalization & mortality during the trial

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No